CLINICAL TRIAL: NCT04795245
Title: J-REGISTER: Japanese REal-world Data for Treatment of Afatinib (GIotrif®) in First-line Setting and Subsequent Therapies for Patients With Advanced EGFR Mutation-positive Lung Adenocarcinoma
Brief Title: Non-interventional Study for Real-world Data of Afatinib Treatment in First-line Setting and of Subsequent Therapies for Patients With Advanced Epidermal Growth Factor Receptor (EGFR) Mutation-positive Lung Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1200-0322
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Non-squamous, Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients treated with afatinib
  Interventions: Drug: afatinib

INTERVENTIONS:
Drug: afatinib — afatinib
  Other Names: Giotrif®

SUMMARY:
The primary objective is to confirm Time on Treatment (TOT) related to afatinib treatment as first-line therapy in patients with Epidermal Growth Factor Receptor (EGFR) mutation-positive Non-Small Cell Lung Cancer (NSCLC).

The observation in the real-world setting of the time from the start of the first-line afatinib until the end of subsequent treatment in this study will provide insights on the sequence of treatment for patients. The Japanese healthcare system will enable this study to evaluate multiple treatment options after afatinib treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Epidermal Growth Factor Receptor (EGFR) mutation-positive advanced Non-Small Cell Lung Cancer (NSCLC)
* Patients who were/are treated with afatinib in the first-line setting at least 20 months* prior to data entry
* Patients 20 years of age or older at the time of consent
* Patients who provided consent to participate in this study (for cases of death or lost to follow-up, instructions from the Ethic Committee (EC)/Institutional Review Board (IRB) at each site should be followed) * Inclusion will be restricted to patients with treatment initiation with afatinib at least 20 months prior to enrolment to avoid early censoring.

Exclusion Criteria:

* Any contraindication to afatinib as specified in the label of Giotrif®
* Patients treated with afatinib within an interventional trial
* Patients with active brain metastases at start of afatinib treatment* * Patients with non-active brain metastases (asymptomatic state) are eligible.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who were treated with afatinib in the first-line setting in each study site after the launch of Giotrif® on 7 May 2014 on a regular basis; their information will be chosen.
  Deceased patients fulfilling the eligibility criteria should be enrolled whenever possible.
Sampling Method: Probability Sample
Enrollment: 805 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nippon Boehringer Ingelheim Co., Ltd., Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Yamaguchi T, Daga H, Tanaka H, Kijima T, Mizushima M. J-REGISTER: real-world study of Japanese patients with EGFR mutation-positive NSCLC treated with first-line afatinib. Future Oncol. 2025 Jul;21(16):2039-2052. doi: 10.1080/14796694.2025.2514423. Epub 2025 Jun 7. PMID 40483538
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Non-interventional, multi-center study from existing data of patients treated with afatinib as the first-line treatment. 40 study sites in Japan were planned for participating. Recruitment of patients was stopped at all sites when it was determined that a sufficient number of patients have been enrolled. A maximum of 50 patients were limited for enrolment per site to avoid differential study site influence on study results. Data extraction started on 01 April 2021 and ended on 07 November 2022.
Pre-assignment Details: Only subjects that met all inclusion and none of the exclusion criteria were included.
Groups:
- Patients Treated With Afatinib: Patients with epidermal growth factor receptor (EGFR) mutation-positive non-small cell lung cancer (NSCLC) treated with afatinib as the first-line treatment during the period from launch of afatinib (7 May 2014) to at least 20 months prior to the time point of enrolment of patients (first round) and follow-up data was extracted for the same patients one year after completion of first round during the study period (second round). Patients were treated with 20, 30, 40 or 50 milligram (mg) tablet of afatinib once daily as indicated in the approved label of afatinib (Giotrif®).
Period: Overall Study
Arm/Group | Patients Treated With Afatinib
Started | 805
Completed (Participants still on afatinib treatment at end of observation period.) | 85
Not Completed | 720
Not completed — Unkown reason | 7
Not completed — Death | 17
Not completed — Other than listed | 19
Not completed — Adverse Event | 143
Not completed — Progressive disease | 512
Not completed — Unknown if patients were still on treatment at end of observation period | 22

BASELINE CHARACTERISTICS:
Population: Final analysis set: All patients who were enrolled in this study and were not excluded due to violations.
Arm/Group | Patients Treated With Afatinib
Number analyzed (Participants) | 805
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.8 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 440
  Male | 365
Race/Ethnicity, Customized [Number; unit: Participants]
  Japanese | 799
  Other Asian | 4
  Non-Asian | 2

OUTCOME MEASURES:

1. Primary Outcome: Time on Treatment (TOT) With Afatinib in First-line TOT (TOT1)
Description: Time on Treatment (TOT) with afatinib in first-line TOT (TOT1). This was assessed as the time from the start of afatinib as first-line treatment until the end of afatinib treatment or death date by any cause, whichever occurs first. If patients did not discontinue first-line treatment with afatinib and did not die at the data extraction, they were censored on the date they were last verified to have been on first-line treatment with afatinib. The survival probability rate (95% confidence interval) against time to first-line treatment failure at 18 months and at 36 months is reported.
Time Frame: From start of afatinib as first line treatment up to 18 months and up to 36 months.
Population: Final analysis set: All patients who were enrolled in this study and were not excluded due to violations.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Patients Treated With Afatinib
Number analyzed (Participants) | 805
Proportion of participants
  At 18 months | 0.39 [0.35 to 0.42]
  At 36 months | 0.15 [0.12 to 0.17]

2. Secondary Outcome: Time on Treatment From the Start of Afatinib Until End of Subsequent Therapies in the Second-line Setting or Death by Any Cause (TOT)
Description: Time on treatment from the start of afatinib until end of subsequent therapies in the second-line setting or death by any cause (TOT). If patients did not discontinue second-line treatment and did not die at the data extraction, they were censored on the date they are last verified to have been on second-line treatment. If patients were on first-line treatment and did not move to second-line treatment at the data extraction, ToT is same as first-line TOT (ToT1) for these patients. The survival probability rate (95% confidence interval) against time to treatment failure at 18 months and at 36 months is reported.
Time Frame: From start of afatinib up to 18 months and up to 36 months.
Population: Final analysis set: All patients who were enrolled in this study and were not excluded due to violations.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Patients Treated With Afatinib
Number analyzed (Participants) | 805
Proportion of participants
  At 18 months | 0.58 [0.54 to 0.61]
  At 36 months | 0.30 [0.27 to 0.34]

3. Secondary Outcome: Time on Treatment From Start of the Second-line Treatment Until End of the Second-line Treatment or Death by Any Cause (TOT2)
Description: Time on treatment from start of the second-line treatment until end of the second-line treatment or death by any cause (TOT2). If patients did not discontinue second-line treatment and did not die at the data extraction, they were censored on the date they are last verified to have been on second-line treatment. The survival probability rate (95% confidence interval) against time to second-line treatment failure at 18 months and at 36 months is reported.
Time Frame: From start of afatinib as second line treatment up to 18 months and up to 36 months.
Population: Final analysis set: All patients who were enrolled in this study and were not excluded due to violations.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Patients Treated With Afatinib
Number analyzed (Participants) | 805
Proportion of participants
  At 18 months | 0.17 [0.14 to 0.20]
  At 36 months | 0.09 [0.07 to 0.12]

4. Secondary Outcome: Overall Survival
Description: If patients did not die at the data extraction, they were censored on the date they are last verified to be alive. The survival probability rate (95% confidence interval) at 18 months and at 36 months is reported.
Time Frame: From start of afatinib up to 18 months and up to 36 months.
Population: Final analysis set: All patients who were enrolled in this study and were not excluded due to violations.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Patients Treated With Afatinib
Number analyzed (Participants) | 805
Proportion of participants
  At 18 months | 0.80 [0.78 to 0.83]
  At 36 months | 0.54 [0.51 to 0.58]

5. Secondary Outcome: Time to Initial Dose Reduction of Afatinib
Description: Time to initial dose reduction of afatinib. If patients did not reduce initial dose of afatinib at the data extraction, they were censored on the date they were last verified to have been on the initial dose of afatinib or increased dose of afatinib. The survival probability rate (95% confidence interval) against time to initial dose reduction of afatinib at 18 months and 36 months is reported.
Time Frame: From start of afatinib up to 18 months and up to 36 months.
Population: Participants included in the full analysis set and who had received afatinib at initial dose of 40 mg.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Patients Treated With Afatinib
Number analyzed (Participants) | 594
Proportion of participants
  At 18 months | 0.22 [0.19 to 0.26]
  At 36 months | 0.20 [0.16 to 0.24]

6. Secondary Outcome: Percentage of Participants With Dose Modifications of Afatinib
Description: Percentage of participants with dose modifications of afatinib.
Time Frame: From start of data extraction until end of data extraction, up to 586 days.
Population: Final analysis set: All patients who were enrolled in this study and were not excluded due to violations.
Measure: Number; unit: Percentage of participants
Arm/Group | Patients Treated With Afatinib
Number analyzed (Participants) | 805
Percentage of participants | 73.7

ADVERSE EVENTS:
Time Frame: Adverse events and deaths were collected for approximately 8.5 years.
Description: Final analysis set: All patients who were enrolled in this study and were not excluded due to violations.
Arm/Group | Patients Treated With Afatinib
All-Cause Mortality (participants affected / at risk) | 486/805
Serious Adverse Events (participants affected / at risk) | 8/805
Other Adverse Events (participants affected / at risk) | 43/805
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Treated With Afatinib (N=805)
Acute myocardial infarction (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Anaphylactic reaction (Immune system disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Treated With Afatinib (N=805)
Nasopharyngitis (Gastrointestinal disorders) | 43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT04795245/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/45/NCT04795245/SAP_001.pdf